CLINICAL TRIAL: NCT01586195
Title: An Open-Label, Multicenter, Phase II Study Of Continuous Oral Zelboraf (Vemurafenib) in Patients With Locally-Advanced, Unresectable, Stage IIIc Or Metastatic Melanoma and Activating Exon 15 BRAF Mutations Other Than V600E
Brief Title: Study Of Zelboraf (Vemurafenib) in Patients With Locally-Advanced, Unresectable, Stage IIIc Or Metastatic Melanoma and Activating Exon 15 BRAF Mutations Other Than V600E
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML27763
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vemurafenib (Experimental): Participants with untreated or previously treated locally advanced, unresectable, Stage IIIc or metastatic melanoma who have an activating exon 15 BRAF mutation other than V600E received vemurafenib 960 milligram (mg) orally twice daily (BID) until disease progression.
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib 960 mg BID
  Other Names: Zelboraf

SUMMARY:
This is an open-label, multicenter, single-agent, phase II study of continuous oral Zelboraf (vemurafenib) in participants with locally-advanced, unresectable, stage IIIc or metastatic melanoma and activating exon 15 BRAF mutations other than V600E.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Histologically-confirmed metastatic melanoma (unresectable Stage IIIc or IV) with an activating BRAF mutation other than V600E, as detected by DNA sequencing of exon 15 performed at a centralized laboratory
* Measurable disease (as defined by RECIST, v1.1)
* Adequate recovery from most recent systemic or local treatment for cancer
* Adequate organ function within 28 days prior to initiation of treatment
* For women of childbearing potential, agreement to the use of two acceptable methods of contraception, including one barrier method, during the study and for 6 months after discontinuation of vemurafenib
* For men with female partners of childbearing potential, agreement to use a latex condom and to advise their female partner to use an additional method of contraception during the study and for 6 months after discontinuation of vemurafenib
* Negative serum pregnancy test within 7 days of commencement of treatment in premenopausal women. Women who are either surgically sterile or have been post-menopausal for at least 1 year are eligible to participate in this study
* Agreement not to donate blood or blood products during the study and for at least 6 months after discontinuation of vemurafenib; for male participants, agreement not to donate sperm during the study and for at least 6 months after discontinuation of vemurafenib
* Signed informed consent form (prior to study entry and before performing any study-related procedures)

Exclusion Criteria:

* Invasive malignancy other than melanoma at the time of enrollment and within 2 years prior to first study drug administration, except for adequately treated (with curative intent) basal or squamous cell carcinoma, in situ carcinoma of the cervix, in situ ductal adenocarcinoma of the breast, in situ prostate cancer, or limited stage bladder cancer or other cancers from which the patient has been disease-free for at least 2 years
* Pregnant or breast-feeding
* Inability to swallow pills
* Concurrent anti-tumor therapy (e.g., chemotherapy, other targeted therapy, radiation therapy, including participation in an experimental drug study)
* Radiation therapy </= 1 week prior to first administration of vemurafenib and stereotactic radiotherapy </= 1 day prior to first administration of vemurafenib
* Prior treatment with a BRAF or MEK inhibitor
* Either a concurrent condition (including medical illness, such as active infection requiring treatment with IV antibiotics or the presence of laboratory abnormalities) or history of a prior condition that places the patient at unacceptable risk if he/she were treated with the study drug or confounds the ability to interpret data from the study
* History of congenital long QT syndrome or a corrected QT (QTc) interval > 450 ms at baseline
* Ongoing cardiac dysrhythmia >/= Grade 2
* Unwillingness to practice effective birth control
* Inability to comply with other requirements of the protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (15):
- United States (15):
  - Arizona Cancer Center, Tucson, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - UCLA School of Medicine; Hematology/Oncology, Los Angeles, California
  - The Angeles Clinic and Research Institute, Santa Monica Office, Santa Monica, California
  - University of Colorado; Anschutz Cancer Pavilion, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University; Winship Cancer Institute, Atlanta, Georgia
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Atlantic Health System, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York
  - Mid Ohio Onc Hematology Inc, Columbus, Ohio
  - UPCI Cancer Institute; Cancer Pavillion, Pittsburgh, Pennsylvania
  - Vanderbilt Univ Medical Ctr, Nashville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vemurafenib
Started | 31
Completed | 5
Not Completed | 26
Not completed — Death | 11
Not completed — Withdrawal of Consent | 5
Not completed — Started new anti-melanoma therapy | 1
Not completed — Reason not specified | 9

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population defined as all enrolled participants who received any amount of study drug.
Groups:
- Vemurafenib: Participants with untreated or previously treated locally advanced, unresectable, Stage IIIc or metastatic melanoma who have an activating exon 15 BRAF mutation other than V600E received vemurafenib 960 mg orally BID until disease progression.
Arm/Group | Vemurafenib
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Rate (BORR)
Description: BORR was assessed by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. BORR was defined as the number of participants whose best overall response was a complete response (CR) or partial response (PR). CR was defined as complete disappearance of all target lesions and non-target disease. PR was defined as a >/=30% decrease under baseline of the sum of diameters of all target lesions. BORR was summarized along with the associated exact 95% confidence interval (CI) using the method of Clopper-Pearson.
Time Frame: Up to 42 months
Population: ITT population defined as all enrolled participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 31
percentage of participants | 22.6 [9.6 to 41.1]

2. Secondary Outcome: Time to BORR
Description: In participants with a confirmed CR or PR, time to BORR was defined as the interval between the date of first treatment and the date of first documentation of confirmed CR or PR (whichever occurred first). BORR was assessed by the investigators according to RECIST v1.1. CR was defined as complete disappearance of all target lesions and non-target disease. PR was defined as a >/=30% decrease under baseline of the sum of diameters of all target lesions. Participants without confirmed CR or PR were censored at the date of last tumor assessment. The time to response was summarized using univariate statistics.
Time Frame: From start of treatment up to first documentation of confirmed CR or PR (up to 42 months)
Population: ITT population defined as all enrolled participants who received any amount of study drug. Participants with a confirmed CR or PR were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 7
months | 1.7 [1.6 to 5.6]

3. Secondary Outcome: Duration of Response
Description: In participants with a confirmed CR or PR, duration of response was defined as the time interval between the date of the earliest qualifying response and the date of progressive disease (PD) or death due to any cause. CR was defined as complete disappearance of all target lesions and non-target disease. PR was defined as a >/=30% decrease under baseline of the sum of diameters of all target lesions. PD was defined as a 20% increase in the sum of the longest diameter of target lesions or the appearance of new lesions and increase of at least 5 mm in the sum of diameters of target lesions. Duration of response was summarized using Kaplan-Meier method.
Time Frame: From date of earliest qualifying response up to date of disease progression or death (up to 42 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 7
months | 10.7 [3.4 to 24.9]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was assessed by the investigators according to RECIST v1.1 and defined as the time interval between the date of the first treatment dose and the date of disease progression or death due to any cause, whichever occurred first. PD was defined as a 20% increase in the sum of the longest diameter of target lesions or the appearance of new lesions and increase of at least 5 mm in the sum of diameters of target lesions. PFS was summarized using Kaplan-Meier method.
Time Frame: From start of treatment up to first documentation of disease progression or death (up to 42 months)
Population: ITT population defined as all enrolled participants who received any amount of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 31
months | 5.5 [1.7 to 26.5]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first treatment to the date of death due to any cause. OS was summarized using Kaplan-Meier method.
Time Frame: Date of first treatment to date of death due to any cause (up to 42 months)
Population: ITT population defined as all enrolled participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 31
months | NA [3.1 to NA] — Median OS and upper limit of 95% confidence interval was not estimiable as they were not reached.

6. Secondary Outcome: Percentage of Participants With 6-Month Survival
Time Frame: Baseline to Month 6
Population: ITT population defined as all enrolled participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 31
percentage of participants | 82.4 [62.6 to 92.3]

7. Secondary Outcome: Percentage of Participants With 12-Month Survival
Time Frame: Baseline to Month 12
Population: ITT population defined as all enrolled participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 31
percentage of participants | 61.6 [40.0 to 77.4]

8. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution.
Time Frame: Up to 42 months
Population: Safety population defined as all enrolled participants who received any amount of vemurafenib on study.
Measure: Number; unit: participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 31
participants | 30

ADVERSE EVENTS:
Time Frame: From the randomization of the first participant to the clinical cutoff date (22 April 2015) (approximately 42 months)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution.
Groups:
- Vemurafenib: Participants received vemurafenib 960 mg orally BID.
Arm/Group | Vemurafenib
Serious Adverse Events (participants affected / at risk) | 13/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=31)
Acute coronary syndrome (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Vasogenic cerebral oedema (Nervous system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=31)
Anaemia (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Vision blurred (Eye disorders) | 3
Dry eye (Eye disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 19
Pyrexia (General disorders) | 4
Chills (General disorders) | 2
Cyst (General disorders) | 2
Mass (General disorders) | 2
Nodule (General disorders) | 2
Bacterial infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Sunburn (Injury, poisoning and procedural complications) | 4
Blood creatinine increased (Investigations) | 5
Weight decreased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 4
Disturbance of attention (Nervous system disorders) | 2
Dysaesthesia (Nervous system disorders) | 2
Hyperaesthesia (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 13
Alopecia (Skin and subcutaneous tissue disorders) | 9
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 9
Actinic keratosis (Skin and subcutaneous tissue disorders) | 6
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 6
Blister (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 2
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.